CLINICAL TRIAL: NCT00026949
Title: Pharmacokinetics of Etoposide in Patients With Breast Cancer Receiving High-Dose Etoposide
Brief Title: Study of Etoposide in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990161; 99-C-0161
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-08

CONDITIONS: Breast Cancer
Keywords: Etoposide; Breast Cancer; Pharmacokinetics
MeSH Terms: conditions — Breast Neoplasms

SUMMARY:
This study will examine how the body handles etoposide, a drug used to treat breast cancer. The knowledge gained may lead to more effective use of the drug with fewer side effects in the future.

Breast cancer patients who are receiving etoposide as part of their treatment may participate in this study. Patients will have 18 blood samples (about a teaspoon or less each) drawn over a 72-hour period during and after their infusion of etoposide. The initial blood samples cannot be taken from the same intravenous line (small tube placed in a vein) used to deliver the etoposide, so a second line may have to be placed temporarily to obtain these samples.

DETAILED DESCRIPTION:
Etoposide is a topoisomerase II inhibitor that has a broad range of anticancer activity at conventional doses (100 mg/m(2) daily x 5 days) and is administered in high doses (greater than 1200 mg/m(2)) as a component of pre-transplant myeloablative chemotherapy regimens. Etoposide pharmacokinetics are linear over a 30-fold dose range, but disposition is highly variable. Etoposide is highly protein bound (95%) to albumin, but protein binding (and therefore free drug concentrations) vary widely in cancer patients. Etoposide is eliminated by metabolism and renal excretion, which may also contribute to the variability. The pharmacokinetics of etoposide will be studied in patients receiving high-dose etoposide as part of their pre-transplant preparative regimen, and pharmacokinetic parameters generated from pharmacokinetic modeling will be correlated with clinical and laboratory characteristics and toxicity in order to develop more rational dosing methods.

ELIGIBILITY:
INCLUSION CRITERIA

Age greater than or equal to 18 years.

Patients with breast cancer who are entered on existing Medicine Branch protocols that include high-dose etoposide.

Must be able to provide informed consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33
Dates: Start 1999-08; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Herzig RH. High-dose etoposide and marrow transplantation. Cancer. 1991 Jan 1;67(1 Suppl):292-8. doi: 10.1002/1097-0142(19910101)67:1+3.0.co;2-7. PMID 1984830
- [Background] Hainsworth JD, Greco FA. Etoposide: twenty years later. Ann Oncol. 1995 Apr;6(4):325-41. doi: 10.1093/oxfordjournals.annonc.a059180. PMID 7619747
- [Background] Pfluger KH, Hahn M, Holz JB, Schmidt L, Kohl P, Fritsch HW, Jungclas H, Havemann K. Pharmacokinetics of etoposide: correlation of pharmacokinetic parameters with clinical conditions. Cancer Chemother Pharmacol. 1993;31(5):350-6. doi: 10.1007/BF00686147. PMID 8431968